CLINICAL TRIAL: NCT01880281
Title: Effect of a Meat Versus Vegetarian Diet in 12 Healthy Volunteers on the Excretion of Alpha-ketoglutarate Measured in 24-hours Urine
Brief Title: Effect of the Diet on Urinary Excretion of Alpha-ketoglutarate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michel Burnier (Other)
Responsible Party: Sponsor-Investigator, Michel Burnier, Professor, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 134/13
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Acid Base Disorder
Keywords: G protein-coupled receptor 99; 2-oxoglutarate receptor 1; alpha-ketoglutarate; urine; pH; acidosis; alkalosis; Healthy volunteers
MeSH Terms: conditions — Acidosis; Alkalosis | interventions — Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meat diet without any vegetables or fruits (Active Comparator): The volunteers will follow a diet of 3 days with at least 400g of meat per day. The 3rd day, the volunteers will do a collect of 24-hour urine.
  The investigational's day, they will receive 50meq of ammonium chlorid over a period of one hour in order to avoid the effect of nausea.
  Interventions: Other: Meat and vegetable diet
- Vegetarian diet without any sources of protein (Active Comparator): The volunteers will follow a diet of 3 days with at least 600g of fruits and vegetables per day without any proteins (animal or vegetal like soybean). The 3rd day, the volunteers will do a collect of 24-hour urine.
  The investigational's day, they will receive 1g of bicarbonate.
  Interventions: Other: Meat and vegetable diet

INTERVENTIONS:
Other: Meat and vegetable diet — After having a diet of 3 days and the investigational's day, the volunteers will have the other diet

SUMMARY:
* The G coupled-protein receptors 99 (GPR99) was discovered in 2002 by Wittenberg et al. and is involved as a metabolic receptor. It has been shown that the natural ligand of GPR99 is an intermediate in the Krebs cycle, alpha-ketoglutarate (aKG). Studies done on rats have shown that aKG is measurable in the blood, freely filtered by the glomerulus and highly reabsorbed in the proximal tubule in metabolic acidosis, while it is not reabsorbed in metabolic alkalosis. No absorption or secretion of aKG intervene between the end of the proximal tubule and the final urine. Thus, having a receptor aKG in the distal tubule creates a paracrine communication with the proximal tubule, informing about the acid-base status of the body and allows adjustment of the urinary excretion of acid or base.
* The hypothesis is that GPR99 is aKG sensor in the distal tubules and allow to report the acid-base status (determined by the metabolic activity of the proximal tubule) of the body to the distal tubule. This can then adapt the urinary excretion of acid or base in the final urine. Acidifying the body by a high meat consumption associated with a test of acidification, the kidney should reduce its aKG excretion and the concentration of this metabolite should be even lower in the urine. And vice versa in the case of alkalizing the body through a vegetarian diet associated with an alkalizing test.
* Twelve healthy omnivorous volunteers will be selected. First inclusion visit includes verification of inclusion/exclusion criteria and signed informed consent. Urine and plasma baseline measurements will be performed and volunteers will meet a dietician. This person will tell them concerning meat and vegetarian diet as well as how to have a diet with 6g of salt per day.Volunteers are then randomized in order to determine which diet they will start first.The first phase will last during 4 days. The diet is followed during 3 days, and a 24-hour urine collection will begin on the third day at 7: 00 am. The fourth day, volunteers will have an investigational's day at the investigation's center after completing their urine collection at home (7:00 am). During the day of investigation, volunteers will give their urine (8: 00 am, corresponding to the baseline urine), and then the "meat" arm will receive a tablet of 50meq of NH4Cl and the "vegetarian" arm will receive a tablet of 1g of NaHC03. Volunteers will stay in the investigation center for 6h. Each hour since 8:00am, a urine sample will be taken, and at 3 hours and 6 hours post-tablet, a blood sample will also be made.This investigational's day will be followed by one to two weeks of treatment washing out. After that, the second phase will begin and will as the first phase excepted that the diet will be inversed.

  5 other healthy vegetarian or vegan volunteers are recruited. Inclusion visit is the same as omnivorous volunteers. Only investigational's day at the investigation's center will be performed (no diet, no urine collection).

ELIGIBILITY:
Inclusion Criteria:

* healthy person
* Age >or= 18, <45
* Caucasian
* Non-smoker
* BMI >or= 18, <25
* normal physical examination
* normal ECG 12 pistes
* systolic blood pressure <or= 139 mmHg and diastolic blood pressure <or= 89 mmHG (after 5 minutes lying, 3 measures a 2-minutes interval, left arm)
* Heart rate <or= 90
* Person can understand the written information and the written consent
* Person gave his/her written consent with date and signature before the start of the study
* Urinary pH > or = 6.5 in the fist urine of the day ( for vegetarian / vegan volunteers only)

Exclusion Criteria:

* vegetarian or vegan diet ( for omnivorous volunteers only)
* electrolytic disorder defined by Na, K, total calcium, phosphate out of the reference's values of laboratory
* seropositive for HIV, HBV or HCV
* Positive for drugs detected in urine (opiates, cannabinoids, cocaine, benzodiazepines, amphetamines, barbiturates)
* fall of systolic or diastolic blood pressure > 10mmHg after one minute standing or all other postural hypotension
* any clinically significant disease or condition at gastrointestinal, respiratory, psychiatric, neurological, renal, hepatic, cardiac and other physical sign abnormality which can interfere with the study
* Pregnant during the screening
* current participation or less than 60 days before the screening to another investigational study
* chronic use of any drug during the 4 weeks preceding the inclusion visit (paracetamol excepted)
* donation of blood, platelets, plasma or bone marrow within 3 months preceding the inclusion visit

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
urinary concentration of alpha-ketoglutarate + plasmatic and urinary pH | up to two investigational's day
  alpha-ketoglutarate measured by titration pH measured by pH-metry

CONTACTS AND LOCATIONS:
Overall Officials: Michel Burnier, professor, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Service de néphrologie, Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Wittenberger T, Hellebrand S, Munck A, Kreienkamp HJ, Schaller HC, Hampe W. GPR99, a new G protein-coupled receptor with homology to a new subgroup of nucleotide receptors. BMC Genomics. 2002 Jul 5;3:17. doi: 10.1186/1471-2164-3-17. Epub 2002 Jul 5. PMID 12098360
- [Background] Gonzalez NS, Communi D, Hannedouche S, Boeynaems JM. The fate of P2Y-related orphan receptors: GPR80/99 and GPR91 are receptors of dicarboxylic acids. Purinergic Signal. 2004 Dec;1(1):17-20. doi: 10.1007/s11302-004-5071-6. PMID 18404396
- [Background] Abbracchio MP, Burnstock G, Boeynaems JM, Barnard EA, Boyer JL, Kennedy C, Miras-Portugal MT, King BF, Gachet C, Jacobson KA, Weisman GA. The recently deorphanized GPR80 (GPR99) proposed to be the P2Y15 receptor is not a genuine P2Y receptor. Trends Pharmacol Sci. 2005 Jan;26(1):8-9. doi: 10.1016/j.tips.2004.10.010. No abstract available. PMID 15629198
- [Background] He W, Miao FJ, Lin DC, Schwandner RT, Wang Z, Gao J, Chen JL, Tian H, Ling L. Citric acid cycle intermediates as ligands for orphan G-protein-coupled receptors. Nature. 2004 May 13;429(6988):188-93. doi: 10.1038/nature02488. PMID 15141213
- [Background] Tokonami N, Morla L, Centeno G, Mordasini D, Ramakrishnan SK, Nikolaeva S, Wagner CA, Bonny O, Houillier P, Doucet A, Firsov D. alpha-Ketoglutarate regulates acid-base balance through an intrarenal paracrine mechanism. J Clin Invest. 2013 Jul;123(7):3166-71. doi: 10.1172/JCI67562. Epub 2013 Jun 24. PMID 23934124